CLINICAL TRIAL: NCT05037305
Title: Knowledge and Attitudes Regarding Pharmacogenetic Testing Among Children With Chronic Conditions and Pregnant Women
Brief Title: VICE-MPRINT: Maternal and Pediatric Pharmacogenetics Survey
Acronym: MPRINT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Digna Velez Edwards, Associate Professor of Pediatrics and Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VUMCIRB:212241
Record Dates: First submitted 2021-08-11; First posted 2021-09-08 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Pharmacogenomic Testing
Keywords: pharmacogenomic; PGx; pediatric; maternal

STUDY DESIGN:
Intervention Model Description: All individuals in study will be undergo pharmacogenetic testing, which will be performed in our CLIA-CAP certified clinical laboratory using the panel-based clinical pharmacogenetic assay used at Vanderbilt University Medical Center. Upon completion of the pharmacogenetic testing, participants will be randomized to view an educational video immediately (intervention group), or after completion of a follow up survey (delayed intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Other): All individuals in the Intervention arm will undergo pharmacogenetic testing, which will be performed in our CLIA-CAP certified clinical laboratory using the panel-based clinical pharmacogenomic assay used at Vanderbilt University Medical Center. Upon completion of the testing, they will be provided a link to an educational video about pharmacogenetic testing and results. Surveys will be performed before and after the pharmacogenetic testing.
  Interventions: Other: Educational video
- Delayed intervention arm (Other): All individuals in the Delayed intervention arm will undergo pharmacogenetic testing, which will be performed in our CLIA-CAP certified clinical laboratory using the panel-based clinical pharmacogenomic assay used at Vanderbilt University Medical Center. Surveys will be performed before and after the pharmacogenetic testing. Upon completion of the first follow up survey, they will be provided a link to an educational video about pharmacogenetic testing and results. A second follow up survey will then be completed.
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — The brief educational video provides information about pharmacogenetic testing, the results of pharmacogenetic testing, and how to find these results in the patient portal.

SUMMARY:
The field of pharmacogenetics has progressed from the discovery of genetic variants that cause variable function of drug metabolism enzymes to a cornerstone of clinical precision medicine. However, there are limited data supporting drug-gene associations for children and for women during and after pregnancy. The unique physiology of childhood and pregnancy demand validation of pharmacogenetic signals prior to clinical implementation. These knowledge gaps are compounded for individuals from minority populations, who have been underrepresented and thus underserved by genomic research and specifically pharmacogenetic studies. The primary objective of this project is to advance research and support clinical implementation in pharmacogenetics for children and pregnant women. This work will illuminate knowledge of, attitudes about, and priorities for pharmacogenetics, and will assess the impact of a brief educational video on knowledge and attitudes around pharmacogenetic testing. The investigators will assess the knowledge and attitudes regarding pharmacogenetic testing among diverse cohorts of children with chronic conditions and pregnant women, before and after receiving pharmacogenetic test results. Participants will be randomized to view an educational video about pharmacogenetic testing either at the time of receiving their pharmacogenetic test results, or at a later time. The investigators will perform surveys before and after pharmacogenomic testing and return of results, and before and after watching the educational video.

DETAILED DESCRIPTION:
This study will follow a two-arm unblinded research design. Study inclusion criteria include ability to provide a DNA sample for pharmacogenetic (PGx) testing and willingness to receive the test results. All participants will have PGx testing. Participants will complete a survey at study baseline, which will collect demographic information (age, race/ethnicity), contact and alternative contact information, primary care physician information, socioeconomic details (e.g. insurance information, education, occupation, marital status, and income) health data (e.g. chronic conditions, personal and family history of genetic diseases) and lifestyle data (e.g. smoking, drinking, and physical activity). Parents will complete enrollment surveys on behalf of children. Basic health and pregnancy history will also be collected for pregnant women. Survey questions regarding information and knowledge on PGx testing will be administered at enrollment and again after return of PGx results. Participants will be randomized to either the intervention group or the delayed intervention group. Individuals in the intervention group will be provided an educational video about PGx testing at the time that PGx results are available. Participants in the Delayed intervention group will be provided the educational video after they complete the first follow up survey. The investigators will include questions in the follow-up survey specific to the educational video in the first follow up survey (Intervention group) or the second follow up survey (Delayed intervention group).

ELIGIBILITY:
Maternal

Inclusion Criteria:

* Provide consent in English or Spanish
* Primary care at VUMC
* Adult women aged 18 and older
* Currently pregnant 12 to 30 weeks gestational age
* Completed or scheduled first prenatal visit at VUMC clinic
* Intent to deliver at VUMC or affiliate
* Agrees to receive findings from pharmacogenomic testing
* Allow access their medical record

Exclusion Criteria:

* Stem cell or solid organ transplant
* Recent transfusion within the previous 2 months
* Inability to provide DNA sample for testing
* Prior pharmacogenomic testing
* Pregnant women undergoing in vitro fertilization or assisted reproductive technologies

Pediatric

Inclusion Criteria:

* Provide consent (parent/guardian) and/or assent (child) in English or Spanish
* Primary care or subspecialty care at VUMC
* Aged 0 to 16
* Parent (0-16 years) and child (12-16 years) agree for both parent and child to receive findings from pharmacogenomic testing
* Parent (0-16 years) and child (12-16 years) allow access their medical record
* Have a chronic health condition.

Exclusion:

* Stem cell or solid organ transplant
* Recent transfusion within the previous 2 months
* Inability to provide DNA sample for testing
* Prior pharmacogenomic testing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Adult pregnant women, and children (regardless of sex)
Enrollment: 500 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Participants' opinions of pharmacogenetic testing changes after results are received | Baseline to post-return of PGx results, approximately 2- 4 weeks
  * Opinion of Knowledge of Pharmacogenetics (PGx) and Related Terminology is being collected in 3 ways. Ten words or phrases will be assessed using a 5-variable ordinal scale ('Not at all familiar' to 'Extremely familiar'). One question will use a 4-variable ordinal scale (Very well, somewhat well, a little, not at all). Another question will use a 5-option Likert scale (A lot, somewhat, a little, not at all, don't know).
  * Opinion of the Usefulness of PGx Testing is being collected using 12 statements with 5-variable ordinal scales ('Strongly disagree' to 'Strongly agree').
  * Opinion of What Can be Learned from PGx Test Results is being collected using 9 statements with 5-variable ordinal scales ('Strongly disagree' to 'Strongly agree').
  For all 3 above, responses reflect relative value, not absolute value, so are not additive and there are no total scores.

SECONDARY OUTCOMES:
Participants gain an improved knowledge of pharmacogenetics after educational intervention | Baseline to post-return of PGx results, approximately 2-4 weeks
  * The 3 sections for Outcome 1 will also be asked to individuals who receive the educational video after they've received their PGx test results (as opposed to those who receive the results and video at the same time). These questions will be used in a pre-post analysis to investigate potential changes in knowledge after receiving the educational intervention.
  * Opinion of the Educational Video: Participants will also be asked questions regarding the video to gauge their perceptions of the utility. These questions are being collected using a 5-variable ordinal scale. There are 4 statements in this section. Response options range from 'Strongly disagree' to 'Strongly agree'. Level of agreement with and understanding of terms is being measured, and responses reflect relative value, not absolute value, so are not additive and there is no total score.
Researchers gain a better understanding of the concerns about and perceptions of pharmacogenetic testing among pregnant women and parents of children with chronic conditions | Baseline to post-return of PGx results, approximately 2- 4 weeks
  * Preferences and Comfort on Their Healthcare Providers Accessing and Using Their PGx Test is assessed using 6 questions with 5-point Likert scales ('Strongly disagree' to 'Strongly agree').
  * Attitudes Regarding PGx Testing and Benefits of the Study are being collected through a matrix block of 12 statements with 5-point Likert scales ('Strongly disagree' to 'Strongly agree').
  * Factors Relating to Decision to Get PGx Testing is measured through a matrix of 8 questions with 5-point Likert scales ('Strongly disagree' to 'Strongly agree').
  * Preference on Provider Who Orders, and Explains PGx Tests will be gauged using 2 "select all that apply" questions.
  * Understanding of, Trust in, and Confidence in Prescriptions after PGx Test Results will be measured with 1 question each.
  For all above, responses reflect relative value, not absolute value, so are not additive and there are no total scores.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets, including genomic data, will be made available upon request and review/approval of research purpose.
Time Frame: It will become available once any manuscripts are accepted for publication. It will be available for a reasonable amount of time.
Access Criteria: Qualified Researchers